CLINICAL TRIAL: NCT06562075
Title: A Post-market-clinical Follow-up Investigation of Safety and Performance by Decoria® Intense Strong
Acronym: DAG-ISJ
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Bohus Biotech AB (Industry)
Collaborators: Key2Compliance (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CIV-24-03-046499
Record Dates: First submitted 2024-08-16; First posted 2024-08-20 (Actual); Last update posted 2025-09-22 (Actual); Status verified 2025-02

CONDITIONS: Jawline Contour Deficit
Keywords: jawline profile

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Investigational Medical Device (Other): All eligable subjects desiring correction of their jawline profile will receive intradermal injection of Decoria Intense Strong on either one or both sides of the face (including or not including the chin).
  Interventions: Device: Decoria Intense Strong

INTERVENTIONS:
Device: Decoria Intense Strong — Decoria® Intense Strong is a HA-based, BDDE-crosslinked dermal filler. Decoria® Intense Strong dermal fillers are injected into dermal tissue to improve and define contouring of jawline profile, supporting overlying tissue to shape facial contours to desired level of correction.
  Appropriate injection volume for the jawline will be determined by the Treating investigator according to IFU

SUMMARY:
A post-market Follow up clinical investigation to confirm the clinical safety and performance profile of Decoria®Intense Strong for the correction and improvement of jawline profile.

DETAILED DESCRIPTION:
This will be a post-market, open label, prospective, interventional, confirmatory, evaluator-blinded,multi - centre, clinical investigation to confirm the clinical safety and performance profile of Decoria®Intense Strong for the correction and improvement of jawline profile.

Subjects desiring correction of their jawline profile at the participating sites will be asked to participate in the clinical investigation. According to national legislation, all subjects must have a consultation with the respective clinic and receive both oral and written information at least 48 hours prior to treatment with fillers, as to allow for sufficient reflection time.

If the subject decides to participate, the subject will receive treatment on Day 0 (Visit 1). At 1 month visit (Visit 2) an optional touch-up may be given as well as assessments performed. All subjects will be followed for 9 months with follow-up and assessments by visits (Visit 2, Visit 3 and Visit 5) and phone call (Visit 4).

Standardized facial photography will be taken prior to and after treatment during Visit 1 and 2 and during each follow-up visit at the clinic (Visit 3 and Visit 5), for evaluation according to GAIS and the exploratory instrumental evaluation of jawline contour. GAIS will be used for blinded-evaluator assessment, treating Investigator assessment and patient satisfaction.

Numeric Pain Rating Scale (NRS) at each visit involving an injection (Visit 1 and Visit 2 - optional touch up) will be used to measure pain.

ELIGIBILITY:
Inclusion Criteria:

1. Adults ≥18 years, males and females.
2. Able and willing to give written informed consent for participation in the investigation.
3. Treating investigator considers the subject's jaw (including or not including chin) amenable to an improvement of at least 1 grade on GAIS. At least one side with either potential to enhance contouring or moderate to severe loss of jawline definition. The grades do not have to be the same on both sides.
4. Ability to follow study instructions and likely to complete all required visits.

Exclusion Criteria:

1. Pregnant or lactating females.
2. Any previous hypersensitivity reaction to any constituent of the Investigational medical device (IMD) or to local anesthetic products.
3. Performed or planned surgery below the nose, permanent implant, injection with fat, and deoxycholic acid that may confound the evaluation of safety and performance of the IMD.
4. Any other intradermal injection, such as semi-permanent fillers or botulinum toxins (no complications are allowed), received in the same injection area within 9 months of the Treatment visit (Visit 1) that may confound the evaluation of safety and performance of the IMD.
5. Has an ongoing episode/relapse, recently diagnosed or newly started medication of an autoimmune disease, as judged by the investigator.
6. Has any chronic or acute skin disease or inflammation (such as pimples, rashes or hives) within or close to the treatment area.
7. Has any treatments (thrombolytics, anticoagulants etc) or disease related to the coagulation system.
8. Subjects that have taken any type of vaccine within two weeks prior injection with the IMD.
9. Patients receiving interferon and ribavirin treatment.
10. Features that may interfere with the visual assessment such as recent cosmetic treatment, scarring, abscess, piercing or tattoo.
11. Participation in a clinical investigation that may affect the safety or performance of this investigation, as judged by the Principal Investigator, or authorized designee.
12. Employees of the study site or the sponsor directly involved with the conduct of the investigation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 110 (Estimated)
Dates: Start 2024-09-06 (Actual); Primary Completion 2025-09 (Estimated); Study Completion 2025-09 (Estimated)

PRIMARY OUTCOMES:
Primary efficacy endpoint | From pre-intervention baseline, at Visit 3 (3 months post baseline).
  The primary efficacy endpoint is the blinded-evaluator assessment of improvement using the Global Aesthetic Improvement Scale (GAIS). GAIS is a comparative scale, based on assessment of change since before pre-intervention, ranges from 1 (exceptional improvement) to 4 (no change) and 5 (worse). The blinded evaluator will compare the pre-intervention face to post-intervention face and assign the level of improvement in the jawline according to the GAIS grading. Each side (left and right) will be assessed independently.
Primary safety endpoint | From baseline to end of study (9 months)
  The primary safety endpoint is to assess the safety of Decoria® Intense Strong, evaluated by the incidence, intensity, duration, and time of onset of related AEs, including injection site reactions, collected during the study duration.

SECONDARY OUTCOMES:
Secondary endpoint | From baseline to visit 2 (1 month optional touch-up)
  1. Pain will be measured by numerical scale Numeric Pain Rating Scale (NRS) (11-point verbal score completed for each target region treated) for each visit involving an injection.
Secondary endpoint | 90 days respectively 270 days after IMD injection
  2. GAIS score at 3 months, and 9 months post-treatment, as assessed by the treating investigator.
Secondary endpoint | 90 days respectively 270 days after IMD injection
  3. GAIS score at 3 months, and 9 months post-treatment, as assessed by the subject.
Secondary endpoint | 30 days between visit 1 and visit 2
  4. Treatment related adverse events and injection site reactions reported after touch-up should be similar to those reported after initial treatment.
Secondary endpoint | 30 days, 90 days and 270 days post-treatment
  5. Change in jawline contour compared to baseline will be measured after treatment, as well as at 1-month, 3-months, and 9-months post-treatment visits.

CONTACTS AND LOCATIONS:
Overall Officials: Lucian Grema, M.D, Principal Investigator — Florakliniken, Stockholm, Sweden
Locations (7):
- Sweden (7):
  - Inskinity, Gothenburg
  - Göteborg Laser & Estetik, Gothenburg
  - Svenska Hudkliniker, Karlstad
  - Inskinity, Stockholm
  - Florakliniken, Stockholm
  - The Faculty, Stockholm
  - Svenska Hudkliniker, Stockholm